CLINICAL TRIAL: NCT03382756
Title: A Cross-over, Randomized and Open-label Clinical Trial to Evaluate the Effects of Food on the Bioavailability of CKD-337 After a Single Oral Dose in Healthy Male Subjects
Brief Title: A Clinical Trial to Assess the Effects of Food on the Bioavailability of CKD-337
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 146FDI17001
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias | interventions — Diet, High-Fat; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Period 1: 1 capsule of test drug(CKD-337) administered under fasting condition
  Period 2: 1 capsule of test drug(CKD-337) under high fat diet condition
  Interventions: Dietary Supplement: High fat diet; Drug: CKD-337
- Group B (Experimental): Period 1: 1 capsule of test drug(CKD-337) under high fat diet fed condition
  Period 2: 1 capsule of test drug (CKD-337) administered under fasting condition
  Interventions: Dietary Supplement: High fat diet; Drug: CKD-337

INTERVENTIONS:
Dietary Supplement: High fat diet — A diet consisting of more than 900kcal and 35% of fat
Drug: CKD-337 — Test Drug
  Other Names: Atorvastatin Calcium Trihydrate + Choline Fenofibrate

SUMMARY:
A cross-over, randomized and open-label clinical trial to evaluate the effects of food on the bioavailability of CKD-337 after a single oral dose in healthy male subjects

DETAILED DESCRIPTION:
This clinical trial is to evaluate the effects of food on pharmacokinetics of CKD-337.

Sixteen male subjects are divided into two groups. A group of subjects are administered a single oral dose of CKD-337 after ingesting high fat meal and the other take same investigational product (IP) in fasting condition. Then their blood is drawn on a fixed schedule to analyse bioavailability of CKD-337.

Finishing the first treatment period, the two groups switch food conditions and initiate the second period. The group of people that were administered CKD-337 with food are then dosed the same IP in fasting condition, and the other group undergo vice versa.

Each treatment period was separated by a washout period of at least 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects between the ages of 19 and 45 years
2. Body mass index between 17.5 and 30.5 kg/m², body weight more than 55kg
3. Subject who doesn't have chronic disease, pathological symptoms or findings
4. Subject who is suitable for the clinical trial determined by laboratory tests(serum test, hematology test, blood chemistry, urinalysis test etc.), Vital Sign, ECG test at the time of screening
5. Subject who fully understand the clinical trial after in-depth explanation, decide to join the clinical trials and sign on an inform consent from willingly.

Exclusion Criteria:

1. Subject who has a clinically significant disease such as hepatic, kidneys, neurological, respiratory, endocrine, hemato-oncology, urinary, cardiovascular, musculoskeletal or psychiatric diseases and who has medical histories listed below.

   * Gallbladder disease including cholelithiasis, severe hepatic impairment
   * Acute/chronic pancreatitis due to hypertriglyceridemia
   * Pulmonary embolism or interstitial lung disease
   * Genetic problems such as galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
   * Hypoalbuminemia
   * Alcoholics
   * Predisposition to rhabdomyolysis
2. Subject who has a history of gastrointestinal disease or gastrointestinal surgery which can affect drug absorption
3. Subject who has hypersensitivity to the drugs containing choline fenofibrate, fenofibrate or atorvastatin, or other drugs such as aspirin, fenofibrate series, antibiotics
4. Subject who has the following clinical significant findings in the EKG at the time of screening

   * QTc(Q-T interval corrected for heart rate) > 450ms
   * PR interval(The interval between the beginning of the P wave and the beginning of the QRS complex in ECG) > 200msec
   * QRS duration(The duration of the QRS wave in ECG) > 120msec
5. Subject whose results of the clinical laboratory tests are included in the following categories

   * CPK(Creatinine Phospho-Kinase) > 2x upper limit of normal range
   * Liver function test (AST;Aspartate Transaminase, ALT;Alanine Transaminase, ALP;Alkaline phosphatase, Total bilirubin, γ-GT;Gamma-Glutamyl Transferase) > 2 x upper limit of normal range
   * eGFR(Estimated Glomerular Filtration Rate) < 60 mL/min/1.73m² Calculated by MDRD(Modification of Diet in Renal Disease)
6. Systolic blood pressure ≥ 160mmHg(millimeter of mercury) or ≤ 100mmHg(millimeter of mercury) , Diastolic blood pressure ≥ 95mmHg(millimeter of mercury) or ≤ 60mmHg(millimeter of mercury) at the time of screening
7. History of drug abuse or a positive reaction for drug abuse examined by urinalysis at the time of screening
8. Subject who took medicines that are known to significantly induce or inhibit drug metabolizing enzymes, including barbiturates, within 30 days prior to the first dose of medication
9. Those who has experienced photoallergy or phototoxicity during treatment with fibrates or ketoprofen
10. Subject who took ETC(Ethical Drug), oriental medicine within 2 weeks and OTC(Over-the-counter Drug), vitamin within 10 days prior to the first dose of medication
11. Subject who took the medication involved in other clinical trials within 3 months prior to the first dose of medication
12. Subject who donated whole conducted blood donation within 2 months or component blood donation or blood transfusion within 1 month prior to the first dose of medication
13. Subject who drinks alcohol more than 21 units per a week (1unit=10g of pure alcohol) continuously within 6 month prior to the first dose of medication or Who can not stop drinking alcohol during the clinical trial
14. Smoker(> 10 cigarettes/day) for the last 3 months or who can not stop smoking during the clinical trial
15. Subject who consumed food containing grapefruit within 48 hours prior to the first dose of medication or who can not stop consumption it until EOS(End of study)
16. Subject who consumed food containing caffeine(e.g. coffee, green tea etc.) within 24 hours prior to the first dose of medication or who can not stop consumption it until discharge
17. Subject who do not use a reliable contraception or who plans a pregnancy during the clinical trial
18. Subject who has unsuitable conditions decided by investigator's judgement including clinical laboratory result

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2017-11-07 (Actual)

PRIMARY OUTCOMES:
AUC0-t of Atorvastatin | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, and 48hr after drug administration
  Area under the plasma concentration of Atorvastatin versus time curve from time zero to time of last quantifiable concentration
Cmax of Atorvastatin | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, and 48hr after drug administration
  Maximum plasma concentration of Atorvastatin
AUCt of Fenofibric acid | Predose(0hr), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, and 96hr after drug administration
  Area under the plasma concentration of Fenofibric acid versus time curve from time zero to time of last quantifiable concentration
Cmax of Fenofibric acid | Predose(0hr), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, and 96hr after drug administration
  Maximum plasma concentration of Fenofibric acid

SECONDARY OUTCOMES:
AUCinf of Atorvastatin | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, and 48hr after drug administration
  Area under the plasma concentration of Atorvastatin versus time curve from time zero to time infinity
Tmax of Atorvastatin | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, and 48hr after drug administration
  Time to maximum concentration of of Atorvastatin
T 1/2 of Atorvastatin | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, and 48hr after drug administration
  Apparent terminal half-life of Atorvastatin
CL/F of Atorvastatin | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, and 48hr after drug administration
  Total body clearance of Atorvastatin
Vd/F of Atorvastatin | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, and 48hr after drug administration
  Apparent volume of distribution of Atorvastatin
AUCinf of Fenofibric acid | Predose(0hr), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, and 96hr after drug administration
  Area under the plasma concentration of Fenofibric acid versus time curve from time zero to time infinity
Tmax of Fenofibric acid | Predose(0hr), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, and 96hr after drug administration
  Time to maximum concentration of Fenofibric acid
T 1/2 of Fenofibric acid | Predose(0hr), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, and 96hr after drug administration
  Apparent terminal half-life of Fenofibric acid
CL/F of Fenofibric acid | Predose(0hr), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, and 96hr after drug administration
  Total body clearance of Fenofibric acid
Vd/F of Fenofibric acid | Predose(0hr), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, and 96hr after drug administration
  Apparent volume of distribution of Fenofibric acid
AUC0-t of 2-hydroxy atorvastatin | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, and 48hr after drug administration
  Area under the plasma concentration of 2-hydroxy atorvastatin versus time curve from time zero to time of last quantifiable concentration
Cmax of 2-hydroxy atorvastatin | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, and 48hr after drug administration
  Maximum concentration attained of 2-hydroxy atorvastatin
AUCinf of 2-hydroxy atorvastatin | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, and 48hr after drug administration
  Area under the plasma concentration of 2-hydroxy atorvastatin versus time curve from time zero to time infinity
Tmax of 2-hydroxy atorvastatin | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, and 48hr after drug administration
  Time to maximum concentration 2-hydroxy atorvastatin
T 1/2 of 2-hydroxy atorvastatin | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, and 48hr after drug administration
  Apparent terminal half-life of 2-hydroxy atorvastatin
CL/F of 2-hydroxy atorvastatin | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, and 48hr after drug administration
  Total body clearance of 2-hydroxy atorvastatin
Vd/F of 2-hydroxy atorvastatin | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, and 48hr after drug administration
  Apparent volume of distribution of 2-hydroxy atorvastatin

CONTACTS AND LOCATIONS:
Overall Officials: Min Kyu Park, Professor, Principal Investigator — Dong-A University Hospital
Locations (1):
- Dong-A University Hospital, Busan, Seo-gu, South Korea